CLINICAL TRIAL: NCT01448876
Title: Time to Cure Chlamydia Trachomatis: Prospective Cohort Study on Detection of Chlamydial RNA and DNA in Anorectal and Cervicovaginal Infections During 8 Weeks After Directly Observed Treatment With Azithromycin
Brief Title: Incubation Time and Test of Cure of Chlamydia Trachomatis
Acronym: Incure
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Incure
Record Dates: First submitted 2011-10-04; First posted 2011-10-07 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2011-10

CONDITIONS: Chlamydia Trachomatis Infection
Keywords: Chlamydia trachomatis; anorectal; cervicovaginal; MSM; women; treatment; RNA; bacterial load; sexual behaviour; Azythromycin treated
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: self-taken cervicovaginal and snorectal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chlamydia care as usual

SUMMARY:
Objective was to understand the dynamics of Chlamydia trachomatis (Ct) detection by nucleic acid amplification testing (NAAT) after treatment and consequences for test-of-cure practice.

DETAILED DESCRIPTION:
Prospective Cohort Study on Detection of Chlamydial ribosomal ribonucleic acid (rRNA) and deoxyribonucleic acid (DNA) in anorectal and cervicovaginal Chlamydia trachomatis (Ct) infections during 8 weeks after directly observed treatment with Azythromycin. The investigators systematically assessed presence of Ct plasmid DNA and rRNA through multiple time-sequential measurements following treatment with 1000mg Azythromycin. By convenience sampling at our outpatient sexually transmitted diseases (STD) clinic, 46 non-pregnant women and 6 men were included, contributing 45 cervicovaginal and 15 anorectal infections. Over a period of 8 weeks, patients provided a total of 1016 self-taken cervicovaginal and/or anorectal swabs (response: 94%). All patients were negative for Human immunodeficiency virus (HIV), gonorrhea and Lymphogranuloma venereum (LGV), tested in anorectal Ct. Usual care was applied by advising abstinence or safe sex for one week and by providing treatment for steady partners. Participants provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Chlamydia trachomatis diagnosis,
* age >=18 years

Exclusion Criteria:

* pregnancy,
* doxycycline treated-Ct,
* recent treatment with antibiotics,
* co-infections with other STD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: By convenience sampling at our outpatient STD clinic, 46 non-pregnant women and 6 men were included, contributing 45 cervicovaginal and 15 anorectal infections.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Duration of detection of Chlamydial rRNA and DNA after treatment | 0 to 52 days after treatment
  At 1,2,3,4,5,6,7,9,12,16,19,23,26,30,37,44, and 52 days post treatment chlamydial rRNA and DNA is measured. Outcomes are the times to rRNA and/or DNA negative test results.

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Service South Limburg, Geleen, South Limburg, Netherlands

REFERENCES:
- [Derived] Dukers-Muijrers NH, Speksnijder AG, Morre SA, Wolffs PF, van der Sande MA, Brink AA, van den Broek IV, Werner MI, Hoebe CJ. Detection of anorectal and cervicovaginal Chlamydia trachomatis infections following azithromycin treatment: prospective cohort study with multiple time-sequential measures of rRNA, DNA, quantitative load and symptoms. PLoS One. 2013 Nov 20;8(11):e81236. doi: 10.1371/journal.pone.0081236. eCollection 2013. PMID 24278400